CLINICAL TRIAL: NCT00591851
Title: Phase II Study of Dose-Dense Doxurubicin and Cyclophosphamide (AC) Followed By Paclitaxel With Trastuzumab in HER2/ NEU-Amplified Breast Cancer: Feasibility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-126
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; adenocarcinoma of the breast; cardiac safety; Breast cancer patients seen at the Memorial Sloan-Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): single arm study
  Interventions: Drug: AC [Adriamycin (A) (also known as doxorubicin) and Cyclophosphamide (C)] Followed By Paclitaxel (P)

INTERVENTIONS:
Drug: AC [Adriamycin (A) (also known as doxorubicin) and Cyclophosphamide (C)] Followed By Paclitaxel (P) — AC [Adriamycin (A) (also known as doxorubicin) and Cyclophosphamide (C)] Followed By Paclitaxel (P)

SUMMARY:
HER-2/neu (+) breast cancer is a more aggressive form of breast cancer. HER-2/neu is a protein that is overproduced by your tumor. It makes your cancer more aggressive. Standard treatments for this type of cancer will help some people, but there is a moderate to high chance that your cancer may come back.

The purpose of this study is to see if a new regimen will be effective in preventing cancer from coming back. This is a phase II trial. In this trial, patient get a drug regimen that has been tested in small groups of people to see what dose is safe. Researchers now wish to see how effective the drug is for HER-2/neu (+) breast cancer. The objective includes looking at short-term side effects and risks of the drug. All of the drugs on this regimen can affect the heart which can be a serious side effect. The drugs affect on heart function is a primary focus.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma breast cancer
* ECOG performance status of 0 or 1
* peripheral neuropathy less than or equal to 1
* discontinued hormonal therapy as a chemoprevention while onstudy
* LVEF by MUGA > 55%?
* Absolute neutrophil count (ANC)> 1000/µL)
* platelet count > 100,000/µL)
* SGOT OR SGPT < 92.5 units/L

Exclusion Criteria:

* Stage IV breast cancer
* any chemotherapy, radiation therapy, immunotherapy, or biotherapy for a CURRENT breast cancer
* pregnant or lactating patients
* active second malignancy, other than adequately treated non-melanoma skin cancers or in situ cervical cancer
* previous allergy/hypersensitivity to Doxorubicin, Cyclophosphamide, Paclitaxel, or other drugs formulated in Cremophor EL?
* unstable angina, congestive heart failure, current use of digitalis, beta-blockers, or calcium blockers for therapy of congestive heart failure, arrhythmia requiring medical therapy, or a history of a myocardial infarction within 12 months
* psychiatric illness that prevents her from understanding the nature of this study and complying with protocol requirements?
* active, unresolved infections
* sensitivity to E. coli derived proteins
* prior chemotherapy with an anthracycline
* prior Herceptin therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chau Dang, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 12/20/2004 Protocol Closed to Accrual 07/25/2006 Primary Completion Date 06/24/2008 Recruitment Location is the medical clinic.
Groups:
- AC Followed by Paclitaxel + Trastuzumab: Doxorubicin and Cyclophosphamide (60/600 mg/m2) X 4 followed by Paclitaxel (175 mg/m2) X 4 every 2 weekly with pegfilgrastim (6mg on day 2) + Trastuzumab x 1 year.
Period: Overall Study
Arm/Group | AC Followed by Paclitaxel + Trastuzumab
Started | 70
Completed | 64
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | AC Followed by Paclitaxel + Trastuzumab
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 49 [27 to 72]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Saftey
Description: LVEF by Muga scan
Time Frame: Baseline-18 months
Measure: Median (Full Range); unit: percentage of LVEF
Arm/Group | AC Followed by Paclitaxel + Trastuzumab
Number analyzed (Participants) | 70
percentage of LVEF
  LVEF at Baseline | 68 [55 to 81]
  LVEF at Month 2 | 67 [58 to 79]
  LVEF at Month 6 (67/70 pts) | 66 [52 to 75]
  LVEF at Month 9 (68/70 pts) | 65 [50 to 75]
  LVEF at Month 18 (48/70 pts) | 66 [57 to 75]

ADVERSE EVENTS:
Arm/Group | AC Followed by Paclitaxel + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 19/70
Other Adverse Events (participants affected / at risk) | 48/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC Followed by Paclitaxel + Trastuzumab (N=70)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Non Cardiac-Chest pain (General disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Fever (General disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC Followed by Paclitaxel + Trastuzumab (N=70)
Alanine aminotransferase increased (Investigations) | 6 (7)
Fatigue (General disorders) | 28 (44)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (17)
Anemia (Blood and lymphatic system disorders) | 19 (43)
White blood cell decreased (Investigations) | 10 (18)
Nausea (Gastrointestinal disorders) | 13 (15)
Neutrophil count decreased (Investigations) | 7 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes